CLINICAL TRIAL: NCT03023527
Title: Nivolumab Role in the Treatment of Patients With Refractory or Relapse Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety
Sponsor: PETHEMA Foundation (Other)
Collaborators: Celgene (Industry); Bristol-Myers Squibb (Industry); Adknoma Health Research, S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM-NIVOPOMDEX
Record Dates: First submitted 2017-01-11; First posted 2017-01-18 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Multiple Myeloma
Keywords: Refractory; Relapsed; Nivolumab
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Nivolumab; pomalidomide; Dexamethasone; elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nivo-pom-dex (Experimental): Nivolumab in combination with Pomalidomide and low dose dexamethasone
  Interventions: Drug: Nivolumab; Drug: Pomalidomide; Drug: Dexamethasone
- nivo-pom-dex-elo (Experimental): Pomalidomide in combination with Nivolumab , dexamethasone and elotuzumab
  Interventions: Drug: Nivolumab; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Elotuzumab

INTERVENTIONS:
Drug: Nivolumab
Drug: Pomalidomide
Drug: Dexamethasone
Drug: Elotuzumab
  Arms: nivo-pom-dex-elo

SUMMARY:
This is an open-label, non-randomized Phase 1 study evaluating the role of two regimens:

A) Nivolumab in combination with Pomalidomide and low dose dexamethasone and B) Nivolumab + Elotuzumab + Pomalidomide + dexamethasone in the treatment of relapse or refractory multiple myeloma patients.

The study will be performed in 10 sites in Spain. First, the MTD for the Nivo-Pom-Dex combination will be determined using a 3+3 scheme. Once the MTD has been determined both Regimes (A and B) will be open for full accrual and patients will be included in an alternating way in both regimes simultaneously. In the case that an unacceptable toxicity was seen in the Lead-in phase (Nivolumab + Pomalidomide + low dose dexamethasone), the other phase would not be open.

A safety analysis by an internal review committee will be performed once the first six patients included in the regimen B have completed the first two cycles.

The main purpose of the study is to analyze the proportion of subjects, with refractory or relapsed multiple myeloma, receiving the combination Nivo-Pom-dex or Nivo-Pom-dex-Elo experience one or more haematological and non haematological SAE (grade 3 or higher).

Additionally, other

Research Hypothesis:

The combination of nivolumab with pomalidomide and dexamethasone will demonstrate adequate safety and tolerability to permit further testing of these combinations in subjects with multiple myeloma. The addition of elotuzumab to nivolumab, pomalidomide and dexamethasone will not change the safety profile.

Duration of Study:

The study will remain open for enrolment for 15 months (estimated), or until the planned total number of 40 subjects is reached if this happens first.

The follow-up of the last recruited patient will be up to 3 years, being the Final analyses performed 1,5 years after the last patient is included.

Study Population:

Male and female adult patients with Multiple Myeloma in first or subsequent relapses, previously exposed to both a proteasome inhibitor and a IMID (Lenalidomide). Patients may be exposed, relapsed or refractory to Lenalidomide.

DETAILED DESCRIPTION:
Test Product, Dose and Mode of Administration, Duration of Treatment:

The study is using a modified 3+3 design and has 2 parts. First (Lead-In phase), the MTD for the Nivo-Pom-dex combination will be determined:

Regimen A: The treatment regimen will include Pomalidomide, Nivolumab and low dose dexamethasone. There will be three different dose levels:

* First dose level (DL1): Nivolumab 240mg intravenous infusion, every other week; Pomalidomide at the standard dose of 4 mg/day from day 1 to 21 in a 28-day cycle and Dexamethasone 40mg weekly except for patients older than 75 or with comorbidities who will received 20 mg weekly.

Initially, 3 patients will be enrolled and treated. If not DLT, 3 additional patients will be included at the same dose level.

* In the case there is DLT, the dose level will be de-escalated.

  * If the DLT is haematological or non-hematological attributable to Pomalidomide, the dose level will be DL-1P (Pomalidomide 2 mg/d from day 1-21, Nivolumab 240mg every other week and Dexamethasone 40mg weekly or 20 weekly in patients older than 75 or with comorbidities.
  * In the case the DLT is non-hematological, and attributable to Nivolumab, this combination arm will be stopped. No Nivolumab dose reductions are allowed in the trial.

Once the MTD has been determined, both regimens A and B will be open for full accrual and patients will be included in an alternating way in both regimens simultaneously.

Regimen B: The treatment regimen will include Pomalidomide and Nivolumab at the selected dose level from the previous arm of the study. Dexamethasone will be given in the standard dose of 40mg weekly on days 1, 8, 15 and 22 of each 28-day cycle and could be reduced to 20mg weekly in case of age above 75 year-old or comorbidities. Elotuzumab will be given at the standard dose of 10mg/kg weekly for the first two cycles, and then on days 1 and 15 for the subsequent cycles.

Treatment will be maintained until disease progression.

Criteria for Evaluation:

* Safety: Adverse events will be assessed continuously during the study and for 100 days after the last treatment. Adverse events will be coded using the most current version of MedDRA and reviewed for potential significance and importance. Adverse events will be evaluated according to the NCI CTCAE Version 4.0. Subjects should be followed until all treatment related adverse events have recovered to grade ≤ 1 or baseline, or are deemed irreversible by the investigator. Safety assessments will be based on medical review of adverse event reports and the results of vital sign measurements, ECGs, physical examinations, and clinical laboratory tests.
* Efficacy: Disease assessment will be performed with serum and urine myeloma lab tests, bone marrow assessment and computed tomography (CT) and/or magnetic resonance imaging (MRI), as appropriate. Myeloma responses will be based on investigator assessment and determined as defined by IMWG criteria. Any initial assessment will be confirmed by a repeat evaluation every 4 weeks.
* Biomarker Assessments: Peripheral blood and bone marrow samples will be collected from subjects to assess mechanisms of primary resistance (cell surface protein analyses and transcriptome analyses) and mechanisms of chemosensitivity to NivoPomDex combination (10-colour flow cytometry, TCR clonality by NGS).

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure nor part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patient must be at least 18 year-old.
* Patient must have a confirmed diagnosis of symptomatic multiple myeloma and measurable secretory disease defined as either serum monoclonal protein of ≥ 0,5 g/dl or urine monoclonal (light chain) protein ≥ 200 mg/24 h. For patients in whom disease is only measurable by serum FLC, the involved FLC should be ≥ 10mg/L (100 mg/dl), with an abnormal serum FLC ratio.
* Patients must have an ECOG performance status of 0, 1 or 2.
* Patient has a multiple myeloma in first or second relapse must be exposed, relapsed or refractory to IMiD (Revlimid) are eligible for the study. Induction therapy followed by autologous stem cell transplantation and consolidations in considered one regimen.
* Patient has the following laboratory values within 14 days before baseline visit (Day 1 Cycle 1 before study drug administration): Platelet count ≥ 75 x 109/L, Haemoglobin ≥ 8.0 g/dl. White blood cell count (WBC) ≥ 2.0 x 109/L, Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; lower values (platelets ≥ 30 x 109/L and neutrophil count (ANC) ≥ 0,5 x 109/L may be accepted if clearly due to heavy bone marrow involvement by multiple myeloma, more than 50% of plasma cell infiltration). Corrected serum calcium < 11.5 mg/dl. Aspartate transaminase (AST) ≤ 3 x upper Total Bilirubin ≤ 1.5 x the upper limit of normal (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL) or ≤ 2 x upper limit normal if Lenalidomide is being prescribed. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min as per Crockoft-Gault formula.
* Women of childbearing potential must be practicing a highly effective method of birth control consistent with local regulations and with the pomalidomide pregnancy prevention plan requirements (see Appendix 5) regarding the use of birth control methods for subjects participating in clinical studies: e.g. established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods: condom with spermicidal foam/gel/film/cream/suppository; male partner sterilization (the vasectomized partner should be the sole partner for that subject); true abstinence (when this is in line with the preferred and usual lifestyle of the subject) during and after the study (6 months after the last dose of any component of the treatment regimen).
* Women of childbearing potential must have two negative pregnancy tests (sensitivity of at least 25 mIU/mL) prior to starting study treatment. The first pregnancy test must be performed within 10-14 days and 24 hours prior to the start of any study drug. Females of childbearing potential with regular or no menstrual cycles must agree to have pregnancy tests weekly for the first 28 days of study participation and then every 28 days while taking the study drug, at study discontinuation, and at day 28 following the last dose of treatment.
* Females of reproductive potential must commit either to abstain continuously from heterosexual sexual intercourse or to use two methods or reliable birth control simultaneously.

Exclusion Criteria:

* Subject has received previous treatment with Nivolumab, Elotuzumab or Pomalidomide.
* Subject has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM) or plasma cell leukemia.
* Subject has previously received autologous stem cell transplantation within 12 weeks before Cycle 1 Day 1, or has received other anti-myeloma treatment within 2 weeks before Cycle 1 Day 1 (with the exception of an emergency use of a short course of corticosteroids (maximum 4 days).
* Subject who had previously received allogeneic stem cell transplantation.
* Subject has peripheral neuropathy or neuropathic pain grade 2 or higher, as defined by the National Cancer Institute Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.
* Prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years. Exceptions include: Basal or squamous cell carcinoma of the skin, Carcinoma in situ of the cervix or breast, incidental histological finding of prostate cancer (TNM stage of T1a or T1b).
* Hypersensitivity to Pomalidomide or Dexamethasone.
* Subjects with any one of the following: congestive heart failure (NYHA class III or IV), myocardial infarction within 2 months prior to starting the study treatment, unstable or poorly controlled angina pectoris (including Prinzmetal variant angina pectoris), known or suspected amyloidosis or arrhythmia.
* Has an active autoimmune disease or a documented history of autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the trial.
* Has a diagnosis of immunosuppressive disorder or is on any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Subject has had radiation therapy within 28 days of Cycle 1 Day 1, except for a localized plasmacytoma, that is not the only evidence of the disease.
* Subject has meningeal involvement of multiple myeloma.
* Subjects unable or unwilling to undergone antithrombotic prophylactic treatment.
* Pregnant or breastfeeding females.
* Known human immunodeficiency virus (HIV) positivity, active infectious hepatitis A, B or C or chronic hepatitis B or C, or any other active infection..
* Incidence of gastrointestinal disease that may significantly alter the absorption of Pomalidomide.
* Subject who received any of the following within the last 21 days of initiation of study treatment: major surgery (except kyphoplasty) or use of any anti-myeloma drug therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Safety of Nivolumab: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 month
  Define Nivolumab DMT in combination with Pomalidomide and dexamethasone at low doses in patients with relapsing MM after one or two treatment lines, and confirm that this DMT is unaffected by the addition of Elotuzumab

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - ICO Badalona, Badalona
  - Hospital Clinic, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Canarias, Las Palmas de Gran Canaria
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Morales Messeguer, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Llatzer, Palma de Mallorca
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Complejo Hospitalario Regional Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miguel JS, Weisel K, Moreau P, Lacy M, Song K, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Belch A, Palumbo A, Schey S, Sonneveld P, Yu X, Sternas L, Jacques C, Zaki M, Dimopoulos M. Pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone alone for patients with relapsed and refractory multiple myeloma (MM-003): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1055-1066. doi: 10.1016/S1470-2045(13)70380-2. Epub 2013 Sep 3. PMID 24007748
- [Background] Chen DS, Irving BA, Hodi FS. Molecular pathways: next-generation immunotherapy--inhibiting programmed death-ligand 1 and programmed death-1. Clin Cancer Res. 2012 Dec 15;18(24):6580-7. doi: 10.1158/1078-0432.CCR-12-1362. Epub 2012 Oct 19. PMID 23087408
- [Background] Topalian SL, Drake CG, Pardoll DM. Targeting the PD-1/B7-H1(PD-L1) pathway to activate anti-tumor immunity. Curr Opin Immunol. 2012 Apr;24(2):207-12. doi: 10.1016/j.coi.2011.12.009. Epub 2012 Jan 9. PMID 22236695
- [Background] Chen DS, Mellman I. Oncology meets immunology: the cancer-immunity cycle. Immunity. 2013 Jul 25;39(1):1-10. doi: 10.1016/j.immuni.2013.07.012. PMID 23890059
- [Background] Fife BT, Bluestone JA. Control of peripheral T-cell tolerance and autoimmunity via the CTLA-4 and PD-1 pathways. Immunol Rev. 2008 Aug;224:166-82. doi: 10.1111/j.1600-065X.2008.00662.x. PMID 18759926
- [Background] Ribas A. Tumor immunotherapy directed at PD-1. N Engl J Med. 2012 Jun 28;366(26):2517-9. doi: 10.1056/NEJMe1205943. Epub 2012 Jun 2. No abstract available. PMID 22658126
- [Background] Brahmer JR. Immune checkpoint blockade: the hope for immunotherapy as a treatment of lung cancer? Semin Oncol. 2014 Feb;41(1):126-32. doi: 10.1053/j.seminoncol.2013.12.014. Epub 2013 Dec 12. PMID 24565586
- [Background] Wang SF, Fouquet S, Chapon M, Salmon H, Regnier F, Labroquere K, Badoual C, Damotte D, Validire P, Maubec E, Delongchamps NB, Cazes A, Gibault L, Garcette M, Dieu-Nosjean MC, Zerbib M, Avril MF, Prevost-Blondel A, Randriamampita C, Trautmann A, Bercovici N. Early T cell signalling is reversibly altered in PD-1+ T lymphocytes infiltrating human tumors. PLoS One. 2011 Mar 7;6(3):e17621. doi: 10.1371/journal.pone.0017621. PMID 21408177
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Konishi J, Yamazaki K, Azuma M, Kinoshita I, Dosaka-Akita H, Nishimura M. B7-H1 expression on non-small cell lung cancer cells and its relationship with tumor-infiltrating lymphocytes and their PD-1 expression. Clin Cancer Res. 2004 Aug 1;10(15):5094-100. doi: 10.1158/1078-0432.CCR-04-0428. PMID 15297412